CLINICAL TRIAL: NCT06846099
Title: A Phase I/Ib Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Efficacy and Indications of Pl3Kα-Selective Inhibitor RP903 (JS105) in Subjects With Advanced Malignancies
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Efficacy and Indications of RP903
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Risen (Suzhou) Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS105-001-I
Record Dates: First submitted 2025-01-19; First posted 2025-02-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer; Cervical Cancer; Endometrial Cancer; Breast Cancer; Solid Tumor Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: once daily on Days 1-28 of each 28-day cycle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- RP903 arm (Experimental): Ia:Participants will receive RP903 in escalating dose levels with starting dose of 50mg, po qd for each 28-day cycle Ib:Participants will receive RP903 with RP2D, po qd for each 28-day cycle
  Interventions: Drug: RP903

INTERVENTIONS:
Drug: RP903 — Ia:RP903 50mg, 100mg, 200mg, 300mg,350mg,or other dose, po qd for each 28-day cycle； Ib: RP903,RP2D,po qd for each 28-day cycle

SUMMARY:
This is an open phase I/Ib clinical study to evaluate the safety, tolerability, pharmacokinetic (PK) profile, and initial efficacy of RP903 in patients with advanced malignancies who have failed standard treatment or have no standard treatment options. The study was divided into two parts: dose escalation and dose extension (Phase Ia) and clinical extension (Phase Ib).

DETAILED DESCRIPTION:
Phase Ia is divided into two phases of dose escalation and dose extension: This part includes dose escalation and dose extension of RP903 single agent to investigate the safety, tolerability, maximum tolerated dose and pharmacokinetic (PK) characteristics of RP903 single agent.

Phase Ib is the clinical indication expansion phase, and the primary purpose of this phase is to evaluate the initial safety and anti-tumor efficacy in a selected indication target population. After determining RP903 monotherapy RP2D in Phase Ia, SMC will select four advanced malignant tumors with PIK3CA mutations (cervical cancer, endometrial cancer, breast cancer, and ovarian cancer) as indications for clinical expansion studies based on phase Ia efficacy, safety, and pharmacokinetic (PK) data. The dose was determined according to the results of the dose escalation phase and the dose extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to provide fresh or archived tumor tissue sample within 3 years
* Ia (dose escalation phase and dose expansion phase):patients with pathologically confirmed advanced Malignant solid tumour who have experienced Treatment failure, are unable to tolerate standard treatment, or have no standard treatment
* Ib: Patients with advanced malignant solid tumours who have PIK3CA activating mutations, experience treatment failure, are intolerant to standard treatment, or have no standard treatment
* Phase Ia: Solid tumour, not limited to specific types; dose expansion phase will prioritize cervix carcinoma, endometrial cancer, ovarian cancer, and breast cancer.
* Phase Ib:Cervix carcinoma (Expanded Cohort 1)：Having received first-line (including Platinum-based chemotherapy ± bevacizumab) or second-line treatment and having disease progression during or after treatment; (recurrence during or within 12 months after neoadjuvant or adjuvant treatment in previous treatment will be regarded as one treatment line)
* Phase Ib:Endometrial cancer (extension cohort 2)：Progression during or after first-line (including platinum) or second-line treatment of advanced or metastatic disease; (recurrence during or within 12 months after neoadjuvant or adjuvant treatment in previous treatment will be considered as one treatment line)；Sarcoma type not included
* Ovarian cancer (expanded cohort 3) (PIK3CA mutation)：
* Ovarian cancer, fallopian tube cancer, or primary peritoneal carcinoma who have experienced treatment failure or are intolerant to at least one line of cytotoxic therapy ± PARP inhibitor; (recurrence during or within 12 months after neoadjuvant or adjuvant therapy will be considered one line of therapy)
* Pathological types include high-grade serous carcinoma, clear cell carcinoma, or Endometrioid carcinoma
* Breast cancer (extension cohort 4) (PIK3CA mutation)：
* Advanced, recurrent and metastatic breast cancer;
* Prior systemic treatment in at least 1 line and no more than 3 lines (patients who have relapsed during or within 12 months after completion of neoadjuvant/adjuvant endocrine therapy will be considered as one line of endocrine therapy)
* At least one measurable lesion as per RECIST v1.1 (except the dose-escalation phase of monotherapy)
* Eastern Cooperative Oncology Group (ECOG) performance status score: 0-1
* Adequate hematologic and organ function

Exclusion Criteria:

* Patients with known allergy to any component of RP903
* Previously treated with PI3K, mTOR or AKT inhibitors
* Systemic anti-tumor therapy within 4 weeks prior to the first dose
* Presence of leptomeningeal or meningeal metastasis, or presence of signs of carcinomatous Meningitis
* Metastases to bone marrow
* Child-Pugh grade B or C
* Active hepatitis B or C
* History of type I Diabetes mellitus，gestational diabetes or uncontrolled type II Diabetes mellitus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Ia:dose-limiting toxicity(DLTs) | 28 days
  Incidence and severity of dose-limiting toxicity (DLTs)
Ia:Adverse Events | 2 years
  Incidence and severity of Adverse Events(AEs) according to NCI-CTCAE
Ia: serious adverse events | 2 years
  Incidence and severity of serious adverse events(SAEs) according to NCI-CTCAE
Ia: Abnormal changes in Laboratory test and other abnormalities | 2 years
  Incidence and severity of abnormal changes in Laboratory test and other tests with clinically significant according to NCI-CTCAE
Ia: MTD | 2 years
  Maximum Tolerated Dose(MTD)
Ia: MAD | 2 years
  Maximum Administrated Dose(MAD)
Ia:RP2D | 2 years
  Recommended Phase II Dose(RP2D)
Ib:objective response rate(ORR); | 2 years
  Efficacy evaluated by the investigator according to RECIST v1.1: objective response rate (ORR);
Ib:AE | 2 years
  Type, frequency, duration, severity and characteristics of Adverse Events (AEs) according to NCI-CTCAE
Ib:SAE | 2 years
  Type, frequency, duration, severity and characteristics of serious adverse events(SAEs) according to NCI-CTCAE

SECONDARY OUTCOMES:
Ia:the concentration of RP903 or its metabolites (if applicable) | 1 years
  the concentration of RP903 or its metabolites (if applicable) in individual subjects at different time points after administration;
Ia:Cmax | 1 years
  peak concentration
Ia:Ctrough | 1 years
  trough concentration
Ia:Tmax | 1 years
  time to peak
Ia:AUC0-t and AUC0-∞ | 1 years
  area under the plasma drug concentration-time curve
Ia:Vd/F | 1 years
  distribution volume
Ia:CL/F | 1 years
  clearance
Ia:t1/2 | 1 years
  half-life
Ia:Rac | 1 years
  cumulative factor
Ia:ORR | 1 years
  objective response rate
Ia:DoR | 1 years
  duration of response
Ia:DCR | 1 years
  disease control rate
Ia:TTR | 1 years
  time to response
Ia:PFS | 1 years
  progression-free survival
Ia:OS | 1 years
  overall survival
Ib:safety:AE | 2 years
  Type, frequency, duration, severity and characteristics of serious adverse events(SAEs) according to NCI-CTCAE
Ib:safety:SAE | 2 years
  Type, frequency, duration, severity and characteristics of serious adverse events(SAEs) according to NCI-CTCAE
Ib:safety:Body temperature | 2 years
  Body temperature changes according to NCI-CTCAE
Ib:safety:pulse | 2 years
  pulse changes according to NCI-CTCAE
Ib:safety:respiratory rate | 2 years
  respiratory rate changes according to NCI-CTCAE
Ib:safety: blood pressure | 2 years
  blood pressure changes according to NCI-CTCAE
Ib:safety:laboratory test | 2 years
  laboratory test changes according to NCI-CTCAE
Ib:safety:heart rate | 2 years
  heart rate changes according to NCI-CTCAE
Ib:safety:QT | 2 years
  QT changes according to NCI-CTCAE
Ib:safety:QTcF | 2 years
  QTcF changes according to NCI-CTCAE
Ib:safety:PR | 2 years
  PR changes according to NCI-CTCAE
Ib:DoR | 1 years
  duration of response
Ib:DCR | 1 years
  disease control rate
Ib:TTR | 1 years
  time to response
Ib:PFS | 1 years
  progression-free survival
Ib:OS | 2 years
  overall survival
Ib:Concentrations of RP903 or its metabolites | 1 years
  Concentrations of RP903 or its metabolites (if applicable) in individual subjects at different time points after dosing.

OTHER OUTCOMES:
blood glucose | 28days
  To explore the relationship between blood glucose levels in peripheral blood and efficacy;
Insulin | 28days
  To explore the relationship between Insulin levels in peripheral blood and efficacy;
C-peptide | 28days
  To explore the relationship between C-peptide levels in peripheral blood and efficacy;
PIK3CA mutation status | 28days
  To explore the correlation between peripheral blood and tumor tissue PIK3CA mutation status in different indications;
peripheral blood PIK3CA mutation | 28days
  To explore the correlation between peripheral blood PIK3CA mutation and efficacy;

CONTACTS AND LOCATIONS:
Locations (23):
- China (23):
  - Beijing Cancer Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Jilin Cancer Hospital, Changchun
  - Jilin University First Hospital, Changchun
  - Sichuan Cancer Hospital, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Fujian Medical University Union Hospital, Fuzhou
  - Sir Run Run Shaw Hospital, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital & Institute, Jinan
  - Affiliated Hospital of Jining Medical College, Jining
  - Linyi Cancer Hospital, Linyi
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Guangxi Medical University Cancer Hospital, Nanning
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Affiliated Cancer Hospital of Fudan University, Shanghai
  - Liaoning Cancer Hospital&Institute, Shenyang
  - Suining Central Hospital, Suining
  - Hubei Cancer Hospital, Wuhan
  - Ceneral Hosipital of Ningxia Medical University, Yinchuan
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No